CLINICAL TRIAL: NCT04541381
Title: The PhOCus Trial: Implementation of Pharmacogenomic Testing in Oncology Care
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: IRB20-0462
Record Dates: First submitted 2020-09-01; First posted 2020-09-09 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: Gastrointestinal Cancer; Head and Neck Cancer; Dihydropyrimidine Dehydrogenase Deficiency; UGT1A1 Gene Mutation; Breast Cancer
Keywords: Pharmacogenomics
MeSH Terms: conditions — Gastrointestinal Neoplasms; Head and Neck Neoplasms; Dihydropyrimidine Dehydrogenase Deficiency; Breast Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Participants assigned to the control group will receive standard chemotherapy without their doctors receiving any genetic information based on the participants' pharmacogenetic results. DNA (Deoxyribonucleic acid) samples for participants in this group will be stored and tested for genotyping six months later after treatment (or earlier if the participant experiences side effects).
- Pharmacogenomics Group (Experimental): Participants enrolled in the pharmacogenomics group will give a DNA (deoxyribonucleic acid) sample for immediate pharmacogenomic genotyping. Once the genotyping results are in, cancer doctors caring for each participant will have immediate access to clinical decision support based on the participant's genetic results and can make dosing decisions/changes to the participant's chemotherapy prescription.
  Interventions: Other: Availability of clinical decision support based on pharmacogenomic results.

INTERVENTIONS:
Other: Availability of clinical decision support based on pharmacogenomic results. — Availability of clinical decision support based on pharmacogenomic results. These results are designed to provide specific dosing information based on the participant's unique genetics/genomics.
  Arms: Pharmacogenomics Group

SUMMARY:
Doctors leading this study hope to find out if giving study participants' genetic information to cancer care providers will help personalize chemotherapy dosing decisions and decrease common chemotherapy side effects. Doctors leading the study will collect genetic information from study participants using pharmacogenomics/genotyping. Pharmacogenomics is the study of how the differences in our genes can affect our unique response to medications.

This is a randomized study, which means that participants in this study will be randomly assigned (as if "by flip of a coin") to one of two different groups: a "pharmacogenomics group" or "control group".

ELIGIBILITY:
Inclusion Criteria Adult patients receiving oncology care at The University of Chicago Medical Center, and for whom treatment with a fluoropyrimidine and/or irinotecan is planned are eligible.

Individuals of all genders, races and ethnic groups are eligible for this trial. There is no bias towards race, sex, or gender in the clinical trial outlined.

Exclusion Criteria

1. Subjects who have previously been exposed to the planned chemotherapy agent at any time (fluoropyrimidine and/or irinotecan).
2. Subjects enrolled in an investigational trial which would preclude dose modifications of fluoropyrimidine and/or irinotecan chemotherapies.
3. Subjects who have undergone, or are being actively considered for, bone marrow, liver or kidney transplantation.
4. Subjects with a history of or active blood cancer (e.g., leukemia).
5. Chronic kidney disease, as defined by glomerular filtration rate (GFR) < 30/mL/min/1.73m2, due to the risk of decreased drug excretion.
6. Liver dysfunction, as defined by the following laboratory values, due to the risk of decreased drug metabolism: Total bilirubin more than 1.5 mg/dL, aspartate Aminotransferase (AST) and alanine transaminase (ALT) more than 2.5 X upper limit of normal*. (*AST and ALT more than 5 X upper limit of normal if hepatic metastases are present).
7. Subjects who have previously or are currently enrolled in another institutional pharmacogenomic genotyping study, or are known to have previously undergone pharmacogenomic genotyping for the gene(s) of interest via another commercial or other means.
8. Inability to understand and give informed consent to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 860 (Estimated)
Dates: Start 2022-02-07 (Actual); Primary Completion 2027-10-01 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Dose Deviation Rate (Co-Primary Endpoint) | 15 months
  To assess the impact of prospective pharmacogenomic testing on dose intensity deviation rate of chemotherapy during the 1st treatment cycle, comparing control vs. pharmacogenomics-guided arms.
Grade 3 or Higher Toxicity (Co-Primary Endpoint) | 5 years
  To determine the degree to which providing oncologists with comprehensive pharmacogenomic information impacts the incidence of Grade 3 or worse toxicities in subjects receiving chemotherapy. Toxicities will be assessed by Common Terminology Criteria for Adverse Events version 5.

SECONDARY OUTCOMES:
Cumulative Chemotherapy Dose Intensity | 5 years.
  Cumulative drug dose intensity received (function of dose and frequency of drug administration).
Response Rate | 5 years.
  Anti-cancer tumor response based on radiographic assessment (complete response, partial response, stable disease, progressive disease), by tumor type and disease setting.
Progression free survival (PFS) | 5 years
  Progression free survival (PFS) by tumor type and disease setting.
Overall Survival | 5 years
  Overall survival (OS) by tumor type and disease setting.

CONTACTS AND LOCATIONS:
Overall Officials: Peter H. O'Donnell, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF